CLINICAL TRIAL: NCT04045444
Title: Physical Activity Level and Cerebral Oxygenation During Gait in Old People
Brief Title: Cerebral Oxygenation During Gait in Elderly
Acronym: OXYSENIOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHRO-2018-11
Record Dates: First submitted 2019-02-21; First posted 2019-08-05 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Cerebral Oxygenation
Keywords: physical activity; cognitive function; elderly; parkinson; muscle oxygenation; gait parameters
MeSH Terms: conditions — Motor Activity | interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- women non active young people (Experimental): women between 18 and 30 years practice less than 1h of physical activity per week
  Interventions: Other: walking; Other: cognitive task
- men non active young people (Experimental): men between 18 and 30 years practice less than 1h of physical activity per week
  Interventions: Other: walking; Other: cognitive task
- women non active old people (Experimental): women between 60 and 85 years practice less than 1h of physical activity per week
  Interventions: Other: walking; Other: cognitive task
- men non active old people (Experimental): men between 60 and 85 years practice less than 1h of physical activity per week
  Interventions: Other: walking; Other: cognitive task
- women active old people (Experimental): women between 60 and 85 years practice at least 3h of physical activity per week
  Interventions: Other: walking; Other: cognitive task
- men active old people (Experimental): men between 60 and 85 years practice at least 3h of physical activity per week
  Interventions: Other: walking; Other: cognitive task
- women with parkinson's disease (Experimental): women between 60 and 85 years presence of the disease according to the criteria of the UK Parkinson Disease Brain Bank
  Interventions: Other: walking; Other: cognitive task
- men with parkinson's disease (Experimental): men between 60 and 85 years presence of the disease according to the criteria of the UK Parkinson Disease Brain Bank
  Interventions: Other: walking; Other: cognitive task

INTERVENTIONS:
Other: walking — Every participants will performed a set of tasks of 2 min. Each task will be separated by a 2 min resting period. The tasks will be walking at 3 km/h, walking while doing the cognitive task, walking at the preferred speed, walking at the preferred speed while doing the cognitive task.
Other: cognitive task — Every participants will performed a set of tasks of 2 min. Each task will be separated by a 2 min resting period. The tasks will be a cognitive task, a control cognitive task.

SUMMARY:
Ageing is accompanied by a cognitive decline altering gait and increasing the risk of falling. Physical activity could reduce this cognitive decline by an improvement in the oxygen supply to the brain. At the moment, the effect of physical activity on brain oxygenation during walking in elderly has never been described. Moreover, the increase in cognitive request during a dual task could lead to an increase in the risk of falling. In this context, the investigators of Orleans's hospital want to examine the effect of the physical activity level of elderly on their brain oxygenation during walking and during a dual task.

Moreover, Parkinson' patients could display an impairment of gait and cognitive function. Attentional task and dual task situation are particularly impaired in this pathology. This is why the investigators of Orleans's hospital want to also examine cerebral activation of these patients during walking and during a dual task.

The hemodynamic cerebral activation will be studied using the near infrared spectroscopy at the level of the prefrontal cortex. This non-invasive technic allows the evaluation of the regional oxyhemoglobin and deoxyhemoglobin variations induced by cerebral activation.

DETAILED DESCRIPTION:
The main aim of the study is to determine the effect of the physical activity level on variations of the pre-frontal oxygenation during walking and during a dual task in elderly. The other aims are to study the effects of age, gender and the Parkinson' disease on variations of the pre-frontal oxygenation during walking and during a dual task in elderly.

For that, 160 participants (females and males) will be included and 8 groups will be constituted (woman and man non active young people, woman and man non active old people, woman and man active old people, woman and man patients with Parkinson's disease).

Every participants will performed a set of 6 tasks of 2 minutes. Each task will be separated by a 2 minutes resting period. The tasks will be a cognitive task, a control cognitive task, walking at 3 kilometers/hour, walking while doing the cognitive task, walking at the preferred speed, walking at the preferred speed while doing the cognitive task.

During the set, prefrontal oxygenation will be measured using the near infrared spectroscopy.

ELIGIBILITY:
Inclusion Criteria:

* men and women non active young people and men and women non active old people : practice less than one hour of physical activity per week
* men and women active old people: practice at least 3 hours of physical activity per week

Non-Inclusion Criteria :

For all subjects:

* Resting electrocardiographic abnormality, Systolic blood pressure >16
* Heart disease, recent and unusual shortness of breath or needing several pillows to sleep at night, effort/rest chest pain, palpitations with effort, history of discomfort with effort
* Respiratory failure
* Disabling rheumatological pathology for walking
* Neuro-progressive disease or sequelae
* Perceptual disorders
* Medication (neuroleptics, psychotropic treatment modifying alertness) potentially having an impact on walking
* Thickness of the skin fold at the vast lateral area greater than 15 mm
* Inability of the volunteer to perform the Random Generation of Numbers task for at least 1 min or frequency of enunciation numbers during the Random Generation of Numbers task > 4/s
* Refusal to sign informed consent

For the young sedentary group (woman and man) and the senior group (woman and man, sedentary and active):

-Subjective health > 3 out of 5

For the senior group (woman and man, sedentary and active):

* Mini-Mental State Evaluation (MMSE) score < 24
* Geriatric Depression Scale (GDS) score > 10

For the Parkinson group (woman and man):

* Presence of a freezing or clinically embarrassing festination (walking disorder)
* Score of Hoehn and Yahr ≥III

Exclusion Criteria:

-Inability of the volunteer to walk on the treadmill at a speed of 3 km/h without assistance (stand at the helm or ask for help)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 117 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
concentration of cerebral oxyhemoglobin | day 1
  The objective is to determine the effect of physical activity level on variations in cerebral oxygenation (combination of concentration of oxyhemoglobin and deoxyhemoglobin) during simple walking and during double task walking in elderly people.
  Cerebral oxygenation will be determined continuously at rest and during walking. She will be measured non-invasively with a near infrared spectrometry system (Oxymon, Artinis Medical system, Netherlands). This system measures the evolution of the concentration of OxyHb and DeoxyHb by measuring the absorption of light into tissues.
  The measurement of cerebral oxygenation will evaluate the hemodynamic response at the regional level during the cognitive task, the simple walking task and the dual task.
concentration of cerebral deoxyhemoglobin | day 1
  The objective is to determine the effect of physical activity level on variations in cerebral oxygenation (combination of concentration of oxyhemoglobin and deoxyhemoglobin) during simple walking and during double task walking in elderly people.
  Cerebral oxygenation will be determined continuously at rest and during walking. She will be measured non-invasively with a near infrared spectrometry system (Oxymon, Artinis Medical system, Netherlands). This system measures the evolution of the concentration of OxyHb and DeoxyHb by measuring the absorption of light into tissues.
  The measurement of cerebral oxygenation will evaluate the hemodynamic response at the regional level during the cognitive task, the simple walking task and the dual task.

SECONDARY OUTCOMES:
concentration of muscular oxyhemoglobin | day 1
  Study the effect of age and gender on muscular oxygenation during the simple walk and during the double task operation.
  This will be measured non invasively with a near infrared spectrometry system (Oxymon, artinis medical system, netherlands)
concentration of muscular deoxyhemoglobin | day 1
  Study the effect of age and gender on muscular oxygenation during the simple walk and during the double task operation.
  This will be measured non invasively with a near infrared spectrometry system (Oxymon, artinis medical system, netherlands)
measurement of cognitive performance using random number generation task | day 1
  This task is for the particpants to state a number between 0 and 9 randomly at the fastest possible frequency by avoiding to state two consécutives digits one after the other (eg not to stay 5 then 6) . this task will be realised during simple walk and double task.
cardiac frequency | day 1
  Study the effect of age and gender on cardiac frequency during the simple walk and during the double task operation
Step width: distance between the middle support point of each foot with optogait system | day 1
  Study the effect of age on walking parameters during the simple walk and during the double task operation
Scale of perceived difficulties for perception of effort | day 1
  This scale consists of 15 steps of ladder associated with verbal information (ranging from extremely easy for 2 to extremely difficult for 14) allowing the subjective descritpion of the difficulty of the task. With this scale the effect of gender on the perception of effort during the simple walk and during the double task will be studied.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal AUZOU, MD, Principal Investigator — CHR orléans
Locations (1):
- CHR Orléans, Orléans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderton BH. Ageing of the brain. Mech Ageing Dev. 2002 Apr;123(7):811-7. doi: 10.1016/s0047-6374(01)00426-2. PMID 11869738
- [Background] Andres P, Van der Linden M. Age-related differences in supervisory attentional system functions. J Gerontol B Psychol Sci Soc Sci. 2000 Nov;55(6):P373-80. doi: 10.1093/geronb/55.6.p373. PMID 11078107
- [Background] Asllani I, Habeck C, Borogovac A, Brown TR, Brickman AM, Stern Y. Separating function from structure in perfusion imaging of the aging brain. Hum Brain Mapp. 2009 Sep;30(9):2927-35. doi: 10.1002/hbm.20719. PMID 19172645
- [Background] Azulay JP, Van Den Brand C, Mestre D, Blin O, Sangla I, Pouget J, Serratrice G. [Automatic motion analysis of gait in patients with Parkinson disease: effects of levodopa and visual stimulations]. Rev Neurol (Paris). 1996 Feb;152(2):128-34. French. PMID 8761620